CLINICAL TRIAL: NCT07337915
Title: Improving Sleep in Midlife Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: American Pistachio Growers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 25-0194
Record Dates: First submitted 2025-12-10; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Poor Sleep Quality
Keywords: Midlife women; Sleep; Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Snack 1 + HeathyHabits1 (Other): Participants in this arm will consume 2 servings of potato chips per day for 30 days. They will also meet once with a study therapist for discussion and suggestions to improve healthy habits (e.g.,diet/nutrition, activity, sleep).
  Interventions: Behavioral: HealthyHabits1; Other: Snack 1
- Snack 2 + HealthyHabits2 (Other): Participants in this arm will consume 2 servings of pistachios for 30 days. They will also meet once with a study therapist for discussion and suggestions to improve sleep habits.
  Interventions: Behavioral: HealthyHabits2; Other: Snack 2
- Snack 2 + HealthyHabits1 (Other): Participants in this arm will consume 2 servings of pistachios per day for 30 days. They will also meet once with a study therapist for discussion and suggestions to improve healthy habits (e.g.,diet/nutrition, activity, sleep).
  Interventions: Behavioral: HealthyHabits1; Other: Snack 2

INTERVENTIONS:
Behavioral: HealthyHabits1 — Participants in this group will be coached in a one hour session with a study therapist how to improve healthy habits (e.g.,diet/nutrition, activity, sleep).
  Arms: Snack 1 + HeathyHabits1; Snack 2 + HealthyHabits1
Behavioral: HealthyHabits2 — Participants in this group will coached in a one hour session by a study therapist on how to improve sleep habits.
  Arms: Snack 2 + HealthyHabits2
Other: Snack 2 — Participants in this group will consume 2 servings of pistachios daily for 30 days
  Arms: Snack 2 + HealthyHabits1; Snack 2 + HealthyHabits2
Other: Snack 1 — Participants in the group will consume 2 servings of potato chips daily for 30 days.
  Arms: Snack 1 + HeathyHabits1

SUMMARY:
This study purpose of this study to see how consuming pistachios and completing a health intervention session a study therapist may improve sleep health in midlife women with poor sleep. Participants in this study will be asked to consume a study snack for about one month, complete a health education session with a study therapist and record information about their sleep. At baseline and after the intervention we will collect information about sleep, alertness, body composition, and blood lipids.

ELIGIBILITY:
Inclusion Criteria:

* All races and ethnic backgrounds
* Between the ages of 45-65 years old
* Women who meet STRAW staging criteria for late peri-menopause (STRAW score of -1) defined as interval of amenorrhea of 60 days OR meet STRAW staging criteria for early post-menopause (STRAW score of +1a, +1b or +1c) defined as >12 months since last menstrual period
* History of poor sleep quality (Pittsburgh Sleep Quality Index score > 5)
* Able and willing to provide informed consent
* Access to an electronic device with teleconferencing capabilities (Teams, etc)
* Willing to consume study intervention
* Fluent (able to read and write) in English

Exclusion Criteria:

* Pregnancy or lactation
* Recent (within the last 3 months) or current use of any prescription or over the counter medications that may impact sleep quality:

  1. including, systemic steroids, anabolic steroids, growth hormone, immunosuppressants, psychotherapy)
  2. recent (within the last 3 months) change in antidepressant medication useage or dosage
* Untreated comorbid sleep disorders that are no known to be responsive to the behavioral interventions: These sleep disorders include but are not limited to narcolepsy, circadian rhythm disorder/shift work, restless leg syndrome, periodic leg movement disorder, obstructive sleep apnea.
* Evidence of recent severe mental health disorders (e.g., suicide attempt or psychiatric hospitalization in past 3 years) that would, in the opinion of the investigator, affect sleep and/or make it difficult for the participant to the investigators instructions.
* Recent (within past 3 years) treated cancer other than basal cell carcinoma
* Current adherence to a weight-loss or weight-gain diet or use of GLP-1 RA medications
* Active or recent (within the past 12 months) alcohol or substance use disorder
* Allergy to study intervention (tree nuts)
* Any other condition or event considered exclusionary by study PI

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) | Baseline, End of intervention period (up to Week 4)
  PSQI is a questionnaire that assesses sleep quality, including both subjective experiences and objective parameters. There are 19 questions that are grouped into 7 components to create a global score. Each component score of the PSQI ranges from 0 to 3, with 3 indicating the greatest dysfunction or disturbance. The seven component scores are then summed to obtain a global PSQI score, which ranges from 0 to 21. Higher scores indicate poorer sleep quality, with a score greater than 5 suggesting significant sleep difficulties.

SECONDARY OUTCOMES:
Change in Seated blood pressure | Baseline, End of intervention period (up to Week 4)
  In-office diastolic and systolic blood pressure will be measured using standard equipment. Blood pressure will be measures in mmHg.
Change in Body Weight | Baseline, End of intervention period (up to Week 4)
  Body Weight will be measured using a standardized scale and reported in kg.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance | Baseline, End of intervention (up to Week 4)
  PROMIS Sleep Disturbance assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. It is an 4-item questionnaire that has participants answer questions about perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep ranked from "not at all" to "always". A higher score indicates more severe sleep issues.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Related Impairment | Baseline, End of intervention period (up to Week 4)
  The PROMIS Sleep Related Impairment questionnaire measures perception of sleepiness during usual awake hours. It is an 4-item questionnaire that has participants answer questions about how sleepiness interfered with their awake-time activities ranked from "not at all" to "always". A higher score indicates greater inference with sleepiness related interference.
Change in 24-h Urinary Melatonin | Baseline, End of intervention period (up to Week 4)
  Participants will collect urine at home for 24 h to be analyzed for urinary output of 6-sulfatoxymelatonin (aMT6s)melatonin, a metabolite of melatonin. Melatonin is a hormone naturally produced by your body as a signal that it is time for sleep.
Change in plasma IL-6 | Baseline, End of intervention period (up to Week 4)
  Plasma IL-6 will be measured using usual laboratory methodology. IL-6 is an inflammatory marker produced by the body. A decrease in IL-6 is considered an improvement.
Change in Psychomotor Vigilance Testing (PVT) | Baseline, End of intervention period (up to Week 4)
  Alertness and attention will be measured using standard 5 minute psychomotor vigilance testing. PVT simply involves responding to a light by pressing a button on a small handheld device.
Change in sleep health measured by RU-SATED | Baseline, End of intervention period (up to Week 4)
  RU-SATED stands for Regularity, Satisfaction, Alertness, Timing, Efficiency, Duration and is a 6-question validated multidimensional sleep health instrument measuring dimensions of sleep health. Participants are asked to rank components of their sleep health over the previous month. Items are each rated on three-point Likert scale from 0 (Rarely / Never) to 2 (Usually / Always), resulting in a total score from 0 to 12. A higher score indicating better sleep health.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue | Baseline, End of Intervention (Up to Week 4)
  The PROMIS Fatigue questionnaire has 8 questions that ask participants on a five point scale of either 'not at all' to very much' or 'never' to 'always' different statements about fatigue and how it impacted their activities of daily living.
Change in visceral fat | Baseline, End of intervention (up to Week 4)
  Visceral fat will be measured using dual x-ray absorptiometry. A greater change in visceral fat is considered good.
Change in sleep latency assessed by actigraphy | Baseline, End of Intervention (Up to Week 4), Post-intervention (Up to Week 5)
  Sleep latency is defined as time period measured from "lights out," or bedtime, to the beginning of sleep. Sleep latency will be assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep. A mean value will be calculated with 7 days of wear. A negative change from Baseline indicates improvement.
Change in sleep latency assessed by sleep diary | Baseline, Post-intervention (Up to Week 5)
  Sleep latency is defined as time period measured from "lights out," or bedtime, to the beginning of sleep. Sleep latency will be recorded by the participant in a diary. A mean value will be calculated with 7 days. A negative change from Baseline indicates improvement.
Change in total sleep time assessed by sleep diary | Baseline, End of intervention (Up to Week 4), Post-intervention (Up to Week 5)
  Total nocturnal sleep time by diary will be calculated as total time in bed (awaking hour - bedtime hour) from which sleep latency was subtracted. Mean value from the past 7 days at each timepoint will be evaluated. A positive change from Baseline indicates improvement.
Change in total sleep time assessed by actigraphy | Baseline, End of Intervention (Up to Week 4), Post-intervention (Up to Week 5)
  Total nocturnal sleep time will be assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep. Total nocturnal sleep time by actigraphy was total time in bed from which sleep latency, nocturnal wake time, and the time from waking up to leaving the bed were subtracted. Mean value from the past 7 days at each timepoint will be evaluated. A positive change from Baseline indicates improvement.
Change in nocturnal awakenings assessed by actigraphy | Baseline, End of Intervention (Up to Week 4), Post-intervention (Up to Week 5)
  The number of nocturnal awakenings will be assessed by actigraphy which is a non-intrusive tool that measures an individual's movement during sleep. Mean value from the past 7 days at each time point will be evaluated. A positive change from Baseline indicates a worsening.
Change in nocturnal awakenings assessed by sleep diary | Baseline, End of Intervention (Up to Week 4), Post-intervention (Up to Week 5)
  The number of nocturnal awakenings will be recorded by the participant in a diary. Mean value from the past 7 days at each timepoint will be evaluated. A negative change from Baseline indicates improvement.
Change in sleep efficiency assessed by actigraphy | Baseline, End of Intervention (Up to Week 4), Post-intervention (Up to Week 5)
  Sleep efficiency is defined is the percentile of total sleep time (TST) to time in bed (TIB), calculated as [(Total sleep time/total time in bed) * 100]. Sleep efficiency will be assessed by actigraphy, a non-intrusive tool that measures an individual's movement during sleep. Mean value from the past 7 days at each timepoint will be evaluated. A positive change from Baseline indicates improvement.
Change daytime activity assessed by actigraphy | Baseline, End of Intervention (Up to Week 4), Post-intervention (Up to Week 5)
  Daytime activity level, as evaluated by the number of footsteps, will be assessed by actigraphy, a non-intrusive tool that measures an individual's movement. Mean value from the past 7 days at each timepoint will be evaluated. A positive change from Baseline indicates improvement.
Change in total cholesterol | Baseline, End of intervention (up to Week 4)
  Total cholesterol will be measured using standard laboratory techniques. A decrease in total cholesterol is considered an improvement
Change in high density lipoprotein (HDL) | Baseline, End of intervention (up to Week 4)
  HDL will be measured from a blood sample using standard laboratory techniques. An increase in HDL is usually considered an improvement.
Change in low density lipoprotein (LDL) | Baseline, End of intervention (up to Week 4)
  LDL will be measured from a blood sample using standard laboratory techniques. An decrease in LDL is usually considered an improvement.
Change in triglycerides | Baseline, End of intervention (up to Week 4)
  Triglycerides will be measured from a blood sample using standard laboratory techniques. A decrease in triglycerides is considered an improvement.

OTHER OUTCOMES:
Energy intake assessed 3-day food record | Baseline
  Participants will be asked to complete a 3-day food record using ASA24. The three day average energy intake will be calculated.
Energy intake assessed by 3-day food record | End of intervention period (up to Week 4)
  Participants will be asked to complete a 3-day food record using ASA24. The three day average energy intake will be calculated.
Satisfaction Survey | End of intervention period (up to Week 4)
  Treatment Satisfaction Scale is a 11-question measure provided after treatment. It measures participants' perceptions on the treatment's effectiveness, benefits, and influence on quality of life (e.g., improvements in work productivity, mood, etc.). Questions are measured on a 5-point Likert scale from Not at all to Very Much (6 questions) and also include 5 open ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Lantz, PhD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified study data that are not designated as restricted use will be made available as public use data to the research community by request to the PIs. Users of the public use data must agree to the Terms of Use, which are designed to protect study participants by limiting data use to scientific research and aggregate statistical reporting, prohibiting attempts to identify study participants, and requiring immediate reporting of any disclosure of study participant identity. Data users also agree not to share or redistribute any data downloads.